CLINICAL TRIAL: NCT02784093
Title: Use of Gastrografin in the Management of Fecal Impaction in Patients With Severe Chronic Constipation: A Double-blinded Randomized Controlled Trial
Brief Title: Use of Gastrografin in the Management of Fecal Impaction in Patients With Severe Chronic Constipation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Jianfeng Gong, Associate professor, Jinling Hospital, China
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Gastrografin-FI
Record Dates: First submitted 2016-05-24; First posted 2016-05-26 (Estimated); Last update posted 2017-08-09 (Actual); Status verified 2017-08

CONDITIONS: Fecal Impaction
Keywords: Chronic Constipation; Fecal impaction; Gastrografin; Randomized Controlled Trial
MeSH Terms: conditions — Fecal Impaction | interventions — Enema

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exposure Group (Experimental): Participants were allocated to receive 100 mL of Gastrograﬁn orally once daily for 6 consecutive days.
  Interventions: Drug: Gastrograﬁn
- Control Group (Placebo Comparator): Participants were allocated to receive enemas twice daily for 6 consecutive days.
  Interventions: Procedure: enemas

INTERVENTIONS:
Drug: Gastrograﬁn
  Arms: Exposure Group
Procedure: enemas
  Arms: Control Group

SUMMARY:
Fecal impaction (FI) is a common cause of lower gastrointestinal tract obstruction, and it is the result of chronic or severe constipation and most commonly found in the elderly population. Gastrografin is a water soluble contrast mediate that could act as an osmotic laxative. It has been shown to confer a therapeutic beneﬁt in adhesive small bowel obstruction (SBO). The investigators speculate that gastrografin administrated orally may be more effective than enema in the treatment of fecal impaction induced intestinal obstruction.

ELIGIBILITY:
Inclusion Criteria:

1. A confirmed presence of fecal impaction diagnosed based on the following conditions: large amount of hard stool (impacted faecaloma) in colon or rectum; abdominal radiography was performed for assessment.
2. Rome III criteria for chronic constipation present for ≥8 weeks.

Exclusion Criteria:

1. Patients with a history of colorectal surgery or an organic cause of constipation; pregnancy.
2. Patients with long-term medical conditions potentially associated with constipation (ie, cystic fibrosis, cerebral palsy, hypothyroidism, spinal and gastric anomalies).
3. Patients with medical or psychiatric illness.
4. Patients with abnormal laboratory data or thyroid function.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
the proportion of patients having successful disimpaction | 6 days
  Successful disimpaction was indicated by the passage of watery stools.
the time when patients having successful disimpaction | 6 days
  Successful disimpaction was indicated by the passage of watery stools.

SECONDARY OUTCOMES:
Wexner constipation score | 6 days
  Severity of constipation symptoms was evaluated according to Wexner constipation scale.
Patient Assessment of Constipation-Symptoms (PAC-SYM) score | 6 days
  Severity of constipation symptoms was evaluated according to PAC-SYM questionnaire.
Patient Assessment of Constipation Quality of Life (PAC-QOL) score | 6 days
  Health-related quality of life was assessed using the trial by the PAC-QOL questionnaire.
adverse events and safety | 6 days

CONTACTS AND LOCATIONS:
Overall Officials: Ning Li, MD, Study Director — Department of Generay Surgery, Jinling hosptal, Medical School of Nanjing University
Locations (1):
- Department of Generay Surgery, Jinling hosptal, Medical School of Nanjing University, Nanjing, Jiangsu, China